CLINICAL TRIAL: NCT06017674
Title: The Effectiveness of Intra-articular Pulsed Radiofrequency in Patients With Painful Knee Osteoarthritis
Brief Title: Intra-articular Pulsed Radiofrequency in Chronic Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Burak Erken, Medical Doctor, Başakşehir Çam & Sakura City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022.03.89
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis; Pain, Chronic
Keywords: intra-articular pulsed radiofrequency; knee osteoarthritis; intra-articular steroid injection
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Chronic Pain | interventions — Steroids

STUDY DESIGN:
Intervention Model Description: Single-center, single-blinded, randomized prospective trial
Who Masked: Investigator
Masking Description: Procedures and evaluations were performed by different practitioners
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Intra-articular Pulsed Radiofrequency and Steroid Injection
  Interventions: Procedure: Intra-articular Pulsed Radiofrequency; Drug: Steroid Injection
- Group 2 (Experimental): Only Intra-articular Steroid Injection
  Interventions: Drug: Steroid Injection

INTERVENTIONS:
Procedure: Intra-articular Pulsed Radiofrequency — A 22-gauge 10 cm radiofrequency cannula with a 10-mm active tip was advanced to the mid-tibiofemoral joint under fluoroscopic guidance. After needle insertion, paresthesia-pain and motor stimulation tests were performed using sensory (50 Hz) and motor (2 Hz, 1 V) stimulation to confirm the absence of stimulation. Intra-articular Pulsed Radiofrequency (IAPRF) was applied at 45 V voltage for 20 ms pulse width for 360 s, followed by a 480 ms silent phase. The tissue temperature was adjusted to not exceed 42°C.
  Arms: Group 1
Drug: Steroid Injection — 8 mg dexamethasone was applied into the tibio-femoral joint with a 22-gauge, 10 cm needle under fluoroscopy.

SUMMARY:
The aim of this study is to investigate the additional effect of Intra-articular Pulsed Radiofrequency (IAPRF) on pain and functional activities in addition to intra-articular steroids in patients with grade II and III knee osteoarthritis.

DETAILED DESCRIPTION:
This randomized controlled trial included patients over 18 years of age with knee pain persisting for more than 3 months and stage II-III knee OA according to the Kellgren-Lawrence scale. The participants were randomized into two groups: the IAPRF + steroid injection (Group 1) and only steroid injection (Group 2) groups. The injections were administered under fluoroscopic guidance in both groups, and the needle was advanced to the midline of the tibiofemoral joint in the anteroposterior and lateral views. Group 1 received 8 mg of intra-articular dexamethasone after IAPRF application for 360 s at 45 V voltage, with the temperature not exceeding 42°C. Group 2 received 8 mg of intra-articular dexamethasone only. Pain intensity and participation in daily activities were evaluated using the numerical rating scale (NRS) and Western Ontario and McMaster Universities arthritis index (WOMAC), respectively, before the procedure and 1, 4, and 12 weeks after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years,
* Having knee pain persisting for more than 3 months due to knee osteoarthritis (OA),
* Kellgren-Lawrence Classification grades II and III OA,
* Giving written and verbal informed consents.

Exclusion Criteria:

* Patients with a history of undergoing knee surgery and/or receiving any intra-articular knee injection within the previous 6 months,
* Having a local or systemic infection or a coagulation disorder,
* Patients who refused to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale | 0, 1, 4 and 12 weeks
  Pain levels before and 1, 4, 12 weeks after the procedure were evaluated with Numeric Rating Scale (NRS). The patients were instructed to score their pain intensity on a scale of 0 to 10, where "0" represents "no pain at all" and "10" represents "worst pain ever possible."

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index | 0, 1, 4 and 12 weeks
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) was used to assess daily living activities at all evaluation points.The WOMAC consists of 24 items on three subscales: pain, stiffness, and physical function. All items were scored on a scale of 0 to 4, where "0" represents none, "1" represents mild, "2" represents moderate, "3" represents severe, and "4" represents extreme. The total score ranges from 0 to 96, with a higher score indicating poorer function in daily living activities.

CONTACTS AND LOCATIONS:
Overall Officials: Burak Erken, MD, Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Başakşehir Cam and Sakura Şehir Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Filippiadis D, Tsochatzis A, Petsatodis E, Galanis S, Velonakis G, Giankoulof C, Kelekis A. Intra-Articular Application of Sluijter-Teixera Poisson Pulsed Radiofrequency in Symptomatic Patients with Knee Osteoarthritis: Focus upon Clinical Efficacy and Safety. Pain Res Manag. 2021 Feb 20;2021:5554631. doi: 10.1155/2021/5554631. eCollection 2021. PMID 34518775
- [Result] Masala S, Fiori R, Raguso M, Morini M, Calabria E, Simonetti G. Pulse-dose radiofrequency for knee osteoartrithis. Cardiovasc Intervent Radiol. 2014 Apr;37(2):482-7. doi: 10.1007/s00270-013-0694-z. Epub 2013 Aug 14. PMID 23942592
- [Result] Karaman H, Tufek A, Kavak GO, Yildirim ZB, Uysal E, Celik F, Kaya S. Intra-articularly applied pulsed radiofrequency can reduce chronic knee pain in patients with osteoarthritis. J Chin Med Assoc. 2011 Aug;74(8):336-40. doi: 10.1016/j.jcma.2011.06.004. Epub 2011 Jul 23. PMID 21872812
- [Result] Sluijter ME, Teixeira A, Serra V, Balogh S, Schianchi P. Intra-articular application of pulsed radiofrequency for arthrogenic pain--report of six cases. Pain Pract. 2008 Jan-Feb;8(1):57-61. doi: 10.1111/j.1533-2500.2007.00172.x. No abstract available. PMID 18211593